CLINICAL TRIAL: NCT00884260
Title: Multi-center, Open Label, Single Arm Study to Assess Efficacy, Safety, Bleeding Pattern and Pharmacokinetics of the Ultra Low Dose Levonorgestrel Intrauterine Contraceptive System (LCS) for a Maximum of 3 Years in Women 18 to 40 Years of Age
Brief Title: GA Levonorgestrel Intrauterine Contraceptive System (LCS) Phase III Study China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91775; MAGIC (Other: company internal); 311966 (Other: company internal)
Record Dates: First submitted 2009-04-16; First posted 2009-04-20 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Contraception
Keywords: Contraception; Intrauterine contraception system

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Levonorgestrel IUS (LCS, BAY86-5028)

INTERVENTIONS:
Drug: Levonorgestrel IUS (LCS, BAY86-5028) — In Vitro release rate: 12µg LNG/24h

SUMMARY:
The purpose of this study is to assess the efficacy, safety, bleeding pattern of low dose LNG (12 mg/ 24 hrs), delivered locally by a new intrauterine contraceptive system suitable for use by women 18 to 40 years of age. In addition, pharmacokinetic assessments will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Has, in the opinion of the investigator, suitable general and uterine conditions for inserting the LCS.
* Normal cervical smear (normal cervical smear within the last six months prior to visit 1 presented in writing can be accepted. The cervical smear should be analyzed and reported according to the Bethesda System.)
* Has clinically normal safety laboratory results (i.e., inside the specified range for inclusion).
* Has regular menstrual cycles (length of cycle 21-35 days) (i.e., endogenous cyclicity without hormonal contraceptive use).

Exclusion Criteria:

* Known or suspected pregnancy or is lactating.
* Vaginal delivery, cesarean delivery, or abortion within 6 weeks prior to visit 2.

Note: Postpartum insertions should be postponed until uterus is fully involuted, however not earlier than 6 weeks after delivery. If involution is substantially delayed, consider waiting until 12 weeks postpartum. In case of a difficult insertion and/or exceptional pain or bleeding during or after insertion, physical examination and ultrasound should be performed immediately to exclude perforation.

* History of ectopic pregnancies. Note: For Korea only: History of ectopic pregnancies or high probability of ectopic gestation.
* Infected abortion within 3 months prior to visit 1. Note: For Korea only: Endometritis after delivery or infected abortion within 3 months prior to visit 1.
* Abnormal uterine bleeding of unknown origin.
* Any genital infection (until successfully treated).
* History of, or current, pelvic inflammatory disease
* Congenital or acquired uterine anomaly.
* Any distortion of the uterine cavity (by e.g., fibroids) likely to cause problems (in the opinion of the investigator) during insertion, retention or removal of the LCS.
* History of, diagnosed or suspected genital malignancy, and untreated cervical dysplasia.
* Current deep venous thrombosis or thrombophlebitis; history of deep venous thrombosis.
* Clinically significant endometrial polyp(s), which, in the opinion of the investigator, will interfere with the assessment of the bleeding profile during the study
* Clinically significant ovarian cyst(s)
* Use of any long-acting injectable sex-hormone preparations within 12 months prior to start of study medication, and if entering subset: any sex-hormone administration within one month prior to start of the study medication.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 918 (Actual)
Dates: Start 2009-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Primary efficacy variable is the occurrence of pregnancy, the Pearl Index (PI) is defined as the number of pregnancies per 100 woman years. | 3 years

SECONDARY OUTCOMES:
LCS expulsion rate | 3 years
Discontinuation rates | 3 years
Adverse events | 3 years
Laboratory tests | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (16):
- Australia (4):
  - Ashfield, New South Wales
  - Herston, Queensland
  - Parkville, Victoria
  - Subiaco, Western Australia
- China (9):
  - Guangzhou, Guangdong
  - Wuhan, Hubei
  - Nanjing, Jiangsu
  - Dalian, Liaoning
  - Jinan, Shandong
  - Chengdu, Sichuan
  - Beijing
  - Chongqing
  - Shanghai
- South Korea (3):
  - Sungnam-si, Gyeonggido
  - Seoul, Korea
  - Seoul